CLINICAL TRIAL: NCT07035405
Title: Colchicine for Secondary Prevention After Ischemic Stroke (CHANCE-3 EX): a Multicenter, Double-blind, Placebo-controlled, Randomized Clinical Trial
Brief Title: Colchicine for Secondary Prevention After Ischemic Stroke (CHANCE-3 EX)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shenzhen Medical Academy of Research and Translation (Unknown)
Responsible Party: Principal Investigator, Yongjun Wang, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHANCE-3 EX
Record Dates: First submitted 2025-06-05; First posted 2025-06-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: stroke; colchicine; secondary prevention
MeSH Terms: conditions — Stroke | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine Group (Experimental): Patients in this arm will receive low-dose colchicine in addition to standard medical care
  Interventions: Drug: Colchicine 0.5 mg
- Placebo Colchicine Group (Placebo Comparator): Patients in this arm will receive placebo colchicine in addition to standard medical care
  Interventions: Drug: Placebo colchicine

INTERVENTIONS:
Drug: Colchicine 0.5 mg — Oral colchicine will be initiated with a dose of 0.5 mg per day.
  Arms: Colchicine Group
Drug: Placebo colchicine — Oral placebo colchicine will be initiated with a dose of 0.5 mg per day.
  Arms: Placebo Colchicine Group

SUMMARY:
The role of colchicine in the secondary prevention of ischemic stroke has not been determinded. This multicenter, randomized, double-blind, placebo-controlled, event-driven clinical trial of CHANCE-3 EX was aimed to assess the efficacy and safety of low-dose colchicine versus placebo on reducing the risk of recurrent ischemic stroke, myocardial infarction and vascular death in patients with minor-to-moderate ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. An age of 18-80 years old
2. Minor-to-moderate ischemic stroke (NIHSS<15 at randomization; confirmed by CT or MRI)
3. Within 7-30 days after the most recent qualifying stroke onset
4. Informed consent signed

Exclusion Criteria:

1. Iatrogenic causes (angioplasty or surgery) of stroke
2. mRS>3 at randomization
3. Known allergy, sensitivity or intolerance to colchicine
4. Inflammatory bowel disease (Crohn's or ulcerative colitis) or chronic diarrhea
5. Symptomatic peripheral neuropathy or pre-existing progressive neuromuscular disease or with creatine kinase (CK) level > 3 times the upper limit of normal as measured within the past 30 days and determined to be non-transient through repeat testing
6. A history of cirrhosis, chronic active hepatitis or severe hepatic disease
7. Impaired hepatic (ALT or AST > three times the upper limit of normal range) or kidney (creatinine exceeding 1.5 times of the upper limit of normal range or eGFR less than 50 ml/min) function at randomization
8. Anemia (haemoglobin <10g/dL), thrombocytopenia (platelet count <100×109/L) or leucopenia (white blood cell count <3×109/L) at randomization
9. Comorbid gout or other indications for colchicine use
10. Active infection at randomization (including respiratory tract infection, urinary tract infection, or gastroenteritis)
11. Requiring chronic immunosuppressant, glucocorticoid, or nonsteroidal anti-inflammatory drugs therapy (except aspirin) during the study
12. Usage of contraindicated medications for colchicine at randomization: moderate or strong CYP3A4 inhibitors (clarithromycin, erythromycin, telithromycin, other macrolide antibiotics, ketoconazole, itraconazole, voriconazole, ritonavir, atazanavir, indinavir, other HIV protease inhibitors, verapamil, diltiazem, quinidine, digoxin, disulfiram, etc) or P-gp inhibitors (cyclosporine)
13. Participating in another clinical trial with an investigational drug or device concurrently or during the last 30 days
14. Women of childbearing age who were not practicing reliable contraception and did not have a documented negative pregnancy test
15. Severe non-cardiovascular comorbidity, active malignant tumors or terminal-stage illnesses, with a life expectancy of less than 2 years
16. Clinically significant drug or alcohol abuse in the past year
17. Any other conditions deemed unsuitable for participation in this study or inability to complete study procedures, including but not limited to mental disorders, cognitive or emotional impairments, or physical conditions that may compromise compliance with study protocols and follow-up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7500 (Estimated)
Dates: Start 2025-07-04 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
First Event of ischemic stroke, myocardial infarction and vascular death | From randomization to occurrence of the first event, with a median follow-up time of 24 months
  The descriptive statistics are the number of participants having at least one of the composites of the primary endpoint.

SECONDARY OUTCOMES:
Ischemic stroke | From randomization to event, with a median follow-up time of 24 months.
  The descriptive statistics are presented as the number of participants having had ischemic stroke.
Myocardial Infarction | From randomization to event, with a median follow-up time of 24 months.
  The descriptive statistics are presented as the number of participants having had myocardial infarction.
Vascular death | From randomization to death, with a median follow-up time of 24 months.
  The descriptive statistics are presented as the number of participants having had a vascular death.
mRS 0-1 at 1 year or ≥1-point improvement in mRS score from baseline to 1 year | At 1 year
  The descriptive statistics are presented as the number of participants having had mRS 0-1 at 1 year or ≥1-point improvement in mRS score from baseline to 1 year.
mRS shift | At 1 year

OTHER OUTCOMES:
Any serious adverse event | Through study completion, a median follow-up time of 24 months.
  The descriptive statistics are presented as the number of serious adverse events.
Adverse events of special interest | Through study completion, a median follow-up time of 24 months.
  The descriptive statistics are presented as the number of adverse events of special interest, including gastrointestinal events (diarrhea, flatulence, nausea, vomiting), infection, impaired hepatic function, moderate or severe impaired renal function, myalgia, myopathy, peripheral neuropathy, myelosuppression, orthostatic hypotension, syncope, rash and alopecia.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including de-identified individual participant data and a data dictionary defining each field in the set, can be made available to other researchers on reasonable request and after signing appropriate data sharing agreements.